CLINICAL TRIAL: NCT05094726
Title: A Comparative Study Between Photobiomodulation and Placebo on Functional Capacity and Fatigability in Post Covid-19 Elderly
Brief Title: Effect of PBM on Functional Capacity and Fatigability in Post Covid-19 Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Elbanna, lecturer at faculty of physical therapy at Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rana H Elbanna
Record Dates: First submitted 2021-10-23; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Post Covid-19 Elderly
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: participants will divided into two equal groups , group A will receive photobiomodulation sessions and group B will receive placebo photobiomodulation
Who Masked: Participant
Masking Description: participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): the participant will received photobiomodulation session.
  Interventions: Radiation: photobiomodulation
- Group B (Placebo Comparator): the participant will received placebo photobiomodulation session.
  Interventions: Other: placebo intervention by photobiomodulation device

INTERVENTIONS:
Radiation: photobiomodulation — Photobiomodulation (PBM) describes the use of red or near-infrared light to stimulate, heal, regenerate, and protect tissue that has either been injured, is degenerating, or else is at risk of dying.
  Arms: Group A
Other: placebo intervention by photobiomodulation device — placebo intervention while the photobiomodulation device is on the off mode
  Arms: Group B

SUMMARY:
Participants had randomly divided into two equal groups. Group (A) which is the study group will receive photobiomodulation session two times per week for four weeks. Group (B) will be the control group that will receive placebo photobiomodulation two times per week for four weeks.

DETAILED DESCRIPTION:
group (A):

1. Each participant will sign a consent form after receiving a detailed explanation about the procedure.
2. submaximal exercise capacity using time up and go test will be assessed.
3. fatigability will be assessed using fatigue assessment scale.
4. hemodynamic variables including; Blood pressure, heart rate, oxygen saturation, maximum oxygen consumption will also be assessed.
5. After one month all the assessment procedure will be repeated again.

r group (B):

1. Each participant will sign a consent form after receiving a detailed explanation about the procedure.
2. submaximal exercise capacity using time up and go test will be assessed.
3. fatigability will be assessed using fatigue assessment scale.
4. hemodynamic variables including; Blood pressure, heart rate, oxygen saturation, maximum oxygen consumption will also be assessed.
5. After one month all the assessment procedure will be repeated again.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 75 years of age
* past history of covid 19 in the last year

Exclusion Criteria:

* ( history of a histologically demonstrated malignant carcinoma , hyperthyreosis , epilepsy, light sensitivity )

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
effect of photobiomodulation on fatigability level | after one month of the trial application
  fatigability level will be assessed using fatigability assesment scale
effect of photobiomodulation on functional capacity level | after one month of the trial application
  functional capacity state will be assessed using submaximal exercise test (time up and go test)

CONTACTS AND LOCATIONS:
Overall Officials: Rana H El Banna, PHD, Principal Investigator — Faculty of physical therapy at Cairo University
Locations (1):
- Al Agouza Outpatient Clinic, Giza, Egypt